CLINICAL TRIAL: NCT04449237
Title: The Mechanism Research of Tinnitus Based on Electroencephalogram and Acoustic Therapy Intervention
Brief Title: Mechanism Research of Tinnitus Based on Electroencephalogram and Acoustic Therapy Intervention
Acronym: EEG-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: sunshan
Record Dates: First submitted 2020-06-16; First posted 2020-06-26 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- volunteer (Other): 40 volunteer will not accept any treatment
  Interventions: Other: music therapy
- patients with unmodified music group (Placebo Comparator): 40 participants in this group will listen to music without any modification
  Interventions: Other: music therapy
- patients with modified tinnitus relieving music (Experimental): 40 participants in this group will listen to the music modified according to the matched dominant tinnitus pitch
  Interventions: Other: music therapy

INTERVENTIONS:
Other: music therapy — music therapy: therapeutic sound according to the frequency and loudness of each patient's tinnitus sound, so as to reduce the tinnitus sound.

SUMMARY:
This project aims to systematically and deeply study the central mechanism of tinnitus using electroencephalogram, and further study the treatment mechanism of tinnitus in combination with sound treatment strategies, so as to provide a research basis for clinical treatment of tinnitus.

DETAILED DESCRIPTION:
Tinnitus is one of the most common auditory disturbances in human. The treatment of tinnitus is always not effective, and the standardized treatment of tinnitus has been lacking. With the development of neuroimaging, neuroelectrophysiology and animal models of tinnitus, the central mechanism of tinnitus has been gradually revealed. The possible mechanisms of tinnitus are the increase of spontaneous discharge rate and synchronization of auditory central neurons caused by hearing deprivation, the change of brain topological structure, the reorganization of auditory cortex, and the disorder of limbic system and auditory central regulation of tinnitus patients. EEG, as an important means to study the cerebral cortex, has become an important technical support for the research on the central mechanism of tinnitus. Changes in activity in auditory brain areas associated with tinnitus have been observed using EEG/ERPs, and non-auditory brain areas such as the limbic system and frontal cortices have also been associated with tinnitus mechanisms. This project aims to systematically and deeply study the central mechanism of tinnitus using electroencephalogram, and further study the treatment mechanism of tinnitus in combination with sound treatment strategies, so as to provide a research basis for clinical treatment of tinnitus.

ELIGIBILITY:
Inclusion Criteria:

1. 18-30 years old, male or female;
2. PTA (0.5,1,2kHz) ≤25dB HL;
3. Tinnitus is a major problem faced by patients (except healthy volunteers);
4. tinnitus course > for 3 months;
5. Healthy, no history of other ear diseases, no history of hearing impairment;
6. There are no other medical, psychological or social problems that need urgent treatment, and no other problems that interfere with tinnitus-related treatment;
7. Voluntary tinnitus treatment, and have enough time to cooperate with treatment.

Exclusion Criteria:

1. Pulsatile tinnitus;
2. Acute tinnitus;
3. Tinnitus is associated with severe hearing loss;
4. Tinnitus accompanied by vertigo;
5. Tinnitus accompanied by headache;
6. Tinnitus is accompanied by somatic symptoms, such as neck pain and temporomandibular joint disorder;
7. Post-traumatic tinnitus;
8. Tinnitus is associated with serious psychiatric complications;

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
electroencephalogram evaluation | From date of randomization, assessed every 3 month, up to 24 month
  latency
electroencephalogram evaluation | From date of randomization, assessed every 3 month, up to 24 month
  peak
electroencephalogram evaluation | From date of randomization, assessed every 3 month, up to 24 month
  amplitude
the loudness of tinnitus | From date of randomization, assessed every 3 month, up to 24 month
  estimated by auditory facility, recorded by unit of dB
the frequency of tinnitus | From date of randomization, assessed every 3 month, up to 24 month
  estimated by auditory facility, recorded by unit of Hz
minimum masking level | From date of randomization, assessed every 3 month, up to 24 month
  the minimum volume to masking tinnitus, recorded by unit of dB
Tinnitus Handicapped Inventory | From date of randomization, assessed every 3 month, up to 24 month
  Tinnitus disability is divided into four levels, the first level:
  0-16 points, no disability; Level 2:18-36, slightly disabled; Level 3:38-56, moderate disability; Level 4:58-100, severe disability.
Hospital Anxiety and Distress Scale | From date of randomization, assessed every 3 month, up to 24 month
  0-7 are asymptomatic; 8 -10 respectively belong to suspicious existence; 11 -21 must exist.

IPD SHARING:
Plan to Share IPD: No